CLINICAL TRIAL: NCT00615108
Title: Safety and Effectiveness of Micardis Tablets Taken Once Daily at 40 mg/Day and 80 mg/Day in Hypertension Patients
Brief Title: Nice Morning- Safety and Efficacy Observational Study of Telmisartan in Hypertensive Patients in Multicenters
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Other Study IDs: 502.519
Record Dates: First submitted 2008-01-31; First posted 2008-02-14 (Estimated); Results first posted 2010-01-26 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purpose of this observational study is to survey the safety and effectiveness of the product under the real condition of usual practice in Taiwanese hypertensive patients. During the 8-week observation, the safety profiles and the clinical evaluation in between doses through blood pressure (BP) measurement for overall effectiveness of telmisartan therapy will be concluded.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female. 2. Aged 20 to 80 years old. 3. Patients meet one of following two criteria:

1. Adult essential hypertensive either newly diagnosed and untreated, or previously treated and uncontrolled patients; sitting blood pressure: systolic blood pressure (BP) > 140 mmHg but < 180 mmHg, and/or diastolic BP > 90 mmHg but < 110 mmHg).
2. Patients who are assessed to benefit from the intake of angiotensin II receptor blocker (ARB) monotherapy or as add-on medication.

Exclusion Criteria:

1. Patients with contraindications to telmisartan use (as per the Micardis® Tablets package insert).
2. Known hypersensitivity to the active ingredient or to any of the excipients of Micardis® Tablets.
3. Any other clinical condition which, in the opinion of the attending physician, would not allow safe administration of the study medications.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hypertension patients
Sampling Method: Non-Probability Sample
Enrollment: 3148 (Actual)
Dates: Start 2006-12; Primary Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (17):
- Taiwan (17):
  - Boehringer Ingelheim Investigator Site, Changhua
  - Boehringer Ingelheim Investigator Site 1, Chiayi City
  - Boehringer Ingelheim Investigator Site 2, Chiayi City
  - Boehringer Ingelheim Investigator Site, Keelung
  - Boehringer Ingelheim Investigator Site, Ksohsiung
  - Boehringer Ingelheim Investigator Site, Miaoli
  - Boehringer Ingelheim Investigator Site 1, Taichung
  - Boehringer Ingelheim Investigator Site 2, Taichung
  - Boehringer Ingelheim Investigator Site 1, Tainan
  - Boehringer Ingelheim Investigator Site 2, Tainan
  - Boehringer Ingelheim Investigator Site 1, Taipei
  - Boehringer Ingelheim Investigator Site 2, Taipei
  - Boehringer Ingelheim Investigator Site 3, Taipei
  - Boehringer Ingelheim Investigator Site 4, Taipei
  - Boehringer Ingelheim Investigator Site 5, Taipei
  - Boehringer Ingelheim Investigator Site 6, Taipei
  - Boehringer Ingelheim Investigator Site 7, Taipei

RESULTS

PARTICIPANT FLOW:
Groups:
- Hypertension Patients: Telmisartan 40mg or 80 mg
Period: Overall Study
Arm/Group | Hypertension Patients
Started | 3148
Completed | 2641
Not Completed | 507
Not completed — Adverse Event | 122
Not completed — Other | 370
Not completed — Lost to Follow-up | 15

BASELINE CHARACTERISTICS:
Arm/Group | Hypertension Patients
Number analyzed (Participants) | 3148
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.04 (12.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1525
  Male | 1623

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Achieving Blood Pressure (BP) Control
Description: BP control was defined as diastolic blood pressure/systolic blood pressure DBP/SBP< 90/140 mm-Hg during observation period. BP is measured every four weeks. The observation period is 8 weeks.
Time Frame: 01-Dec-2006 to 31-Dec-2008
Population: Subjects include those who took 20mg, 40mg, 80mg and unknown dosage
Measure: Number; unit: Percentage of Participants
Groups:
- Micardis 40mg: Telmisartan 40 mg
- Micardis 80mg: Telmisartan 80 mg
- Total: Telmisartan 40mg or 80 mg
Arm/Group | Micardis 40mg | Micardis 80mg | Total
Number analyzed (Participants) | 2406 | 205 | 2641
Percentage of Participants | 66 | 46 | 65

2. Secondary Outcome: Percentage of Patients Achieving BP Response
Description: Achieving BP response was defined as reduction from baseline in sitting SBP or DBP > 10 mmHg during the observational period. The observation period is 8 weeks.
Time Frame: 01-Dec-2006 to 31-Dec-2008
Population: Included the patients who took 20mg, 40mg, 80mg and unknown dosage.
Measure: Number; unit: percentage of participants
Arm/Group | Micardis 40mg | Micardis 80mg | Total
Number analyzed (Participants) | 2406 | 205 | 2641
percentage of participants
  Achieving SBP > 10 mmHg | 63 | 63 | 63
  Achieving DBP > 10 mmHg | 40 | 31 | 39

3. Secondary Outcome: Overall Assessment by Patients
Description: Overall assessment was reported as a 5-point scale rated from 0 to 4 as below:
  4: Outstanding 3: Very satisfactory 2: Satisfactory
  1: Marginal 0: Not satisfactory
Time Frame: 01-Dec-2006 to 31-Dec-2008
Population: Included the patients who took 20mg, 40mg, 80mg and unknown dosage.
Measure: Number; unit: Percentage of Participants
Arm/Group | Micardis 40mg | Micardis 80mg | Total
Number analyzed (Participants) | 2512 | 207 | 2791
Percentage of Participants
  Outstanding | 8 | 14 | 8
  Very satisfactory | 34 | 25 | 33
  Satisfatory | 47 | 43 | 47
  Marginal | 9 | 18 | 10
  Not satisfactory | 2 | 8 | 3

4. Secondary Outcome: Overall Assessment by Attending Physicians
Description: as for outcome 3
Time Frame: 01-Dec-2006 to 31-Dec-2008
Population: Included the patients who took 20mg, 40mg, 80mg and unknown dosage
Measure: Number; unit: Percentage of Participants
Arm/Group | Micardis 40mg | Micardis 80mg | Total
Number analyzed (Participants) | 2512 | 207 | 2791
Percentage of Participants
  Outstanding | 10 | 6 | 9
  Very satisfactory | 34 | 24 | 33
  Satisfactory | 45 | 38 | 44
  Marginal | 9 | 22 | 10
  Not satisfactory | 3 | 11 | 4

ADVERSE EVENTS:
Time Frame: 8 Weeks
Arm/Group | Hypertension Patients
Serious Adverse Events (participants affected / at risk) | 16/3148
Other Adverse Events (participants affected / at risk) | 0/3148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hypertension Patients (N=3148)
Vomiting (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Dizziness, Dizzling (Nervous system disorders) | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Hiatus hernia (Gastrointestinal disorders) | 1
Tendon rupture (Musculoskeletal and connective tissue disorders) | 1
Ischaemic cerebral infarction (Vascular disorders) | 1
Ileal ulcer perforation (Gastrointestinal disorders) | 1
Peritonitis (Skin and subcutaneous tissue disorders) | 2
Septic shock (Immune system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Hypertension (Vascular disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1
Hypovolemic shock (Blood and lymphatic system disorders) | 1
Sudden cardiac death (Cardiac disorders) | 1
Subdural haematoma (Blood and lymphatic system disorders) | 1
Haemorrhage (Vascular disorders) | 1
Subarachnoid haemorrhage (Vascular disorders) | 1
Skull fracture (Musculoskeletal and connective tissue disorders) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Chest discomfort (General disorders) | 1
Acute coronary syndrome (Cardiac disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.